CLINICAL TRIAL: NCT02058355
Title: Development and Evaluation of Effectiveness of an Internet-based Brief Intervention for Alcohol Use Among Brazilian College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, André Bedendo, MSc, Federal University of São Paulo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: PNFBrAB2013
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Personalized Normative Feedback (Experimental): This group receive the complete Personalized Normative Feedback (with normative information and a list of consequences)
  Interventions: Behavioral: Consequences List Feedback; Behavioral: Personalized Normative Feedback
- Normative Feedback (Experimental): This group receive a feedback only with normative informations (without a list of consequences)
  Interventions: Behavioral: Personalized Normative Feedback
- Consequences List Feedback (Experimental): This group receive a list of consequences without normative informations
  Interventions: Behavioral: Consequences List Feedback

INTERVENTIONS:
Behavioral: Consequences List Feedback
  Arms: Consequences List Feedback; Personalized Normative Feedback
Behavioral: Personalized Normative Feedback
  Arms: Normative Feedback; Personalized Normative Feedback

SUMMARY:
This project aims to develop and evaluate the effectiveness of an Personalized Normative Feedback (PNF) intervention via the internet, through a randomized clinical trial for alcohol consumption among Brazilian college students, as well as evaluating the most effective components of the PNF (normative and list of consequences). The sample is composed of college students aged between 18 and 30 years. Participants allocated into four different groups: control, full intervention (PNF), feedback with normative components (FN) and feedback with list of consequences (FLC). The investigators will use the dismantling design to study the most effective components. Participants will be followed-up at 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* College students
* Age 18-30 years
* Alcohol Use during the last 3 months

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46142 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Alcohol Consumption | Last 3 Months
  Measured by AUDIT questionnaire

SECONDARY OUTCOMES:
Maximum Drinks | Last 3 months
  Maximum number of drinks reported
Frequency of Alcohol Use | Last 3 months
  Measured by AUDIT questionnaire
Typical Number of Drinks | Last 3 months
  Measured by AUDIT questionnaire
Number of Alcohol-related Consequences | Last 3 Months
  Measured by AUDIT questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, Brazil